CLINICAL TRIAL: NCT02814136
Title: Comparison of Wide Area Circular Ablation With Extra-wide Area Circular Ablation in Subjects With Persistent Atrial Fibrillation, a Randomized Study
Brief Title: Wide Area Circular Ablation Versus Extra-wide Area Circular Ablation in Persistent Atrial Fibrillation
Acronym: WACAvsEWACA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mosaic Life Care (Other)
Responsible Party: Principal Investigator, Mazda Biria, Principle Investigator, Mosaic Life Care
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MLC001
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WACA (Active Comparator): wide area circular ablation
  Interventions: Procedure: Ablation
- EWACA (Active Comparator): extra-wide area circular ablation
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation

SUMMARY:
Ablation of atrial fibrillation is an established method for treatment of subjects with atrial fibrillation with goal of restoration of sinus rhythm. Among different methods, wide area circular ablation (WACA) is shown to provide the same results with fewer complications. This project will compare WACA with extra-wide area circular ablation (E-WACA) in subjects who are considered for ablation of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with symptomatic persistent atrial fibrillation who are scheduled for clinically indicated ablation of AF.

Exclusion Criteria:

* Subjects younger than 18 year of age.
* Subjects who are pregnant.
* Subjects who are unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the achievement of sinus rhythm in subjects undergoing ablation of atrial fibrillation using WACA compared to E-WACA. | 1 year

SECONDARY OUTCOMES:
ii. To compare the time to reoccurrence of atrial fibrillation, atrial flutter and/or atrial tachycardia in subjects undergoing ablation of atrial fibrillation using WACA compared to E-WACA. | 1 year

OTHER OUTCOMES:
iii. To assess the frequency of complications in subjects undergoing ablation of atrial fibrillation using WACA compare to E-WACA. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mazda Biria, MD, Principal Investigator — Physician of Cardiology and Electrophysiology
Locations (1):
- Mosaic Life Care, Saint Joseph, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumagai K, Ogawa M, Noguchi H, Yasuda T, Nakashima H, Saku K. Electrophysiologic properties of pulmonary veins assessed using a multielectrode basket catheter. J Am Coll Cardiol. 2004 Jun 16;43(12):2281-9. doi: 10.1016/j.jacc.2004.01.051. PMID 15193694
- [Background] Jongbloed MR, Schalij MJ, Poelmann RE, Blom NA, Fekkes ML, Wang Z, Fishman GI, Gittenberger-De Groot AC. Embryonic conduction tissue: a spatial correlation with adult arrhythmogenic areas. J Cardiovasc Electrophysiol. 2004 Mar;15(3):349-55. doi: 10.1046/j.1540-8167.2004.03487.x. PMID 15030427
- [Background] Perez-Lugones A, McMahon JT, Ratliff NB, Saliba WI, Schweikert RA, Marrouche NF, Saad EB, Navia JL, McCarthy PM, Tchou P, Gillinov AM, Natale A. Evidence of specialized conduction cells in human pulmonary veins of patients with atrial fibrillation. J Cardiovasc Electrophysiol. 2003 Aug;14(8):803-9. doi: 10.1046/j.1540-8167.2003.03075.x. PMID 12890038
- [Background] Vaitkevicius R, Saburkina I, Rysevaite K, Vaitkeviciene I, Pauziene N, Zaliunas R, Schauerte P, Jalife J, Pauza DH. Nerve supply of the human pulmonary veins: an anatomical study. Heart Rhythm. 2009 Feb;6(2):221-8. doi: 10.1016/j.hrthm.2008.10.027. Epub 2008 Oct 22. PMID 19187915
- [Background] Ouyang F, Bansch D, Ernst S, Schaumann A, Hachiya H, Chen M, Chun J, Falk P, Khanedani A, Antz M, Kuck KH. Complete isolation of left atrium surrounding the pulmonary veins: new insights from the double-Lasso technique in paroxysmal atrial fibrillation. Circulation. 2004 Oct 12;110(15):2090-6. doi: 10.1161/01.CIR.0000144459.37455.EE. Epub 2004 Oct 4. PMID 15466640
- [Background] Pappone C, Rosanio S, Augello G, Gallus G, Vicedomini G, Mazzone P, Gulletta S, Gugliotta F, Pappone A, Santinelli V, Tortoriello V, Sala S, Zangrillo A, Crescenzi G, Benussi S, Alfieri O. Mortality, morbidity, and quality of life after circumferential pulmonary vein ablation for atrial fibrillation: outcomes from a controlled nonrandomized long-term study. J Am Coll Cardiol. 2003 Jul 16;42(2):185-97. doi: 10.1016/s0735-1097(03)00577-1. PMID 12875749
- [Background] Pappone C, Santinelli V, Manguso F, Vicedomini G, Gugliotta F, Augello G, Mazzone P, Tortoriello V, Landoni G, Zangrillo A, Lang C, Tomita T, Mesas C, Mastella E, Alfieri O. Pulmonary vein denervation enhances long-term benefit after circumferential ablation for paroxysmal atrial fibrillation. Circulation. 2004 Jan 27;109(3):327-34. doi: 10.1161/01.CIR.0000112641.16340.C7. Epub 2004 Jan 5. PMID 14707026
- [Background] Arentz T, Weber R, Burkle G, Herrera C, Blum T, Stockinger J, Minners J, Neumann FJ, Kalusche D. Small or large isolation areas around the pulmonary veins for the treatment of atrial fibrillation? Results from a prospective randomized study. Circulation. 2007 Jun 19;115(24):3057-63. doi: 10.1161/CIRCULATIONAHA.107.690578. Epub 2007 Jun 11. PMID 17562956
- [Background] Chae S, Oral H, Good E, Dey S, Wimmer A, Crawford T, Wells D, Sarrazin JF, Chalfoun N, Kuhne M, Fortino J, Huether E, Lemerand T, Pelosi F, Bogun F, Morady F, Chugh A. Atrial tachycardia after circumferential pulmonary vein ablation of atrial fibrillation: mechanistic insights, results of catheter ablation, and risk factors for recurrence. J Am Coll Cardiol. 2007 Oct 30;50(18):1781-7. doi: 10.1016/j.jacc.2007.07.044. Epub 2007 Oct 15. PMID 17964043
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D; Heart Rhythm Society Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. 2012 HRS/EHRA/ECAS expert consensus statement on catheter and surgical ablation of atrial fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design: a report of the Heart Rhythm Society (HRS) Task Force on Catheter and Surgical Ablation of Atrial Fibrillation. Developed in partnership with the European Heart Rhythm Association (EHRA), a registered branch of the European Society of Cardiology (ESC) and the European Cardiac Arrhythmia Society (ECAS); and in collaboration with the American College of Cardiology (ACC), American Heart Association (AHA), the Asia Pacific Heart Rhythm Society (APHRS), and the Society of Thoracic Surgeons (STS). Endorsed by the governing bodies of the American College of Cardiology Foundation, the American Heart Association, the European Cardiac Arrhythmia Society, the European Heart Rhythm Association, the Society of Thoracic Surgeons, the Asia Pacific Heart Rhythm Society, and the Heart Rhythm Society. Heart Rhythm. 2012 Apr;9(4):632-696.
- [Background] Tamborero D, Mont L, Berruezo A, Matiello M, Benito B, Sitges M, Vidal B, de Caralt TM, Perea RJ, Vatasescu R, Brugada J. Left atrial posterior wall isolation does not improve the outcome of circumferential pulmonary vein ablation for atrial fibrillation: a prospective randomized study. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):35-40. doi: 10.1161/CIRCEP.108.797944. Epub 2008 Dec 3. PMID 19808442